CLINICAL TRIAL: NCT02138799
Title: A Phase I, Randomized, Open-label, 2-arm Parallel-design Study to Determine the Effect of Multiple-dose Rifampin on the Pharmacokinetics, Safety and Tolerability of Single-dose Enzalutamide in Healthy Male Subjects
Brief Title: A Study to Evaluate How a Drug That Alters Liver Enzymes (Rifampin) Affects the Metabolism of Enzalutamide in Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9785-CL-0405; 2012-004841-34 (EudraCT Number)
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Drug-Drug Interaction (DDI); Healthy Subjects; Pharmacokinetics of Enzalutamide
Keywords: Phase I; Pharmacokinetics; Safety; Drug-drug interactions; Enzalutamide; Rifampin; CYP3A4; CYP2D8; Enzyme induction
MeSH Terms: interventions — enzalutamide; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: single dose of enzalutamide (Experimental)
  Interventions: Drug: enzalutamide
- 2: multiple doses of rifampin and single dose of enzalutamide (Experimental)
  Interventions: Drug: enzalutamide; Drug: rifampin

INTERVENTIONS:
Drug: enzalutamide — oral
  Other Names: ASP9785,; MDV3100,; Xtandi
Drug: rifampin — oral
  Arms: 2: multiple doses of rifampin and single dose of enzalutamide

SUMMARY:
This study evaluates how a drug that alters liver enzymes (rifampin) affects the metabolism of enzalutamide in men by measuring concentrations of enzalutamide and its metabolites in plasma.

DETAILED DESCRIPTION:
The study consists of 2 randomized treatment arms. In both arms the subjects receive a single oral dose of enzalutamide.

In Arm 1 the subjects are admitted to the clinic on Day -1 where they remain until Day 3. Each subject receives a single oral dose of enzalutamide, administered under fasted conditions on Day 1. Ambulant visits take place from Day 4 to Day 50. Full PK profiles are obtained for enzalutamide, Major Inactive Carboxylic Acid Metabolite (M1) and Active Metabolite N-desmethyl Enzalutamide (M2) from Day 1 up to Day 50 after intake of enzalutamide.

In Arm 2 each subject receives a once-daily dose of rifampin on Days 1 to 21. On Day 8, a single oral dose of enzalutamide is administered under fasted conditions concomitantly with rifampin. Full PK profiles are obtained for enzalutamide, M1 and M2 from Day 8 up to Day 57 after intake of enzalutamide.

An End of Study Visit (ESV) takes place between 7 and 10 days after the last PK sample or early withdrawal.

Safety assessments are performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a Body Mass Index (BMI) of at least 18.5 and no greater than 29.9 kg/m2 at screening.
* Subject must use a condom when having sex with a pregnant woman.
* Male subject and their female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of two forms of birth control.
* Male subject must not donate sperm starting at screening and throughout the study period and for 90 days after the final study drug administration.

Exclusion Criteria:

* Subject has a confirmed CYP2C8 poor metabolizer status based on genotyping analysis.
* Subject has a history of seizure or any condition that may predispose to seizure. Historically or currently on any convulsive medication or drugs that may lower the seizure threshold. History of any central nervous system (CNS) infections. Also history of transient ischemic attack or cerebrovascular accident with or without head trauma within 12 months of enrollment (Day -1 visit).
* Subject has any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission on Day -1.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
PK of enzalutamide and the sum of enzalutamide + M2 in plasma measured by area under the curve (AUC) from time 0 to 336 hours after dosing (AUC0-336h) | Days 1 to 50 (29 times)
PK of enzalutamide and the sum of enzalutamide + M2 in plasma measured by AUC extrapolated to infinity (AUCinf) | Days 1 to 50 (29 times)

SECONDARY OUTCOMES:
PK of enzalutamide, M2, M1 and the sum of enzalutamide + M2 in plasma | Days 8 to 57 (49 times)
  AUC0-336h, AUCinf, Cmax (M2, M1), time to attain Cmax (tmax), terminal elimination half life (t1/2), AUC up to last quantifiable concentration (AUClast), apparent total body clearance after extra vascular dosing (CL/F), apparent volume of distribution during the terminal phase after extra vascular dosing (Vz/F) (parent compound only), Metabolite-to-Parent Ratio (MPR), percent extrapolated for AUCinf (%AUC)
PK of rifampin in plasma | Days 6 to 21 (20 times)
  Cmax, tmax, AUC for the defined interval between doses (AUCtau), minimum concentration (Cmin)
Safety and tolerability of enzalutamide, alone or in the presence of rifampin | Screening (Day -28 to -7) to End of Study Visit (ESV) (>34 times)
  vital signs, incidence of adverse events (AE), laboratory assessments, physical examination, electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Parexel International GmbH, Berlin, Germany